CLINICAL TRIAL: NCT04950452
Title: Exercise Training to Promote Resilience to Chronic Lymphocytic Leukemia in Older Adults by Enhancing Physical and Immunological Reserve
Brief Title: Exercise Training to Promote Resilience to Chronic Lymphocytic Leukemia
Acronym: HIIT-CLL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00094597
Record Dates: First submitted 2021-06-23; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Aging; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLL-EX (Experimental): Subjects will undergo supervised exercise training 3 x per week for 12 weeks. Three/sessions per week will consist of intervals of high-intensity (~85% of maximal capacity) will be 5 to 10 bouts of 30 seconds at this intensity with rest periods in between intervals that range from 30 seconds to 2 minutes. Following this, on 2 occasions/week subjects will complete muscular endurance resistance training on machine weights.
  Interventions: Behavioral: Exercise Training
- CLL-CON (No Intervention): Subjects will not receive supervised exercise training and will be asked to maintain their daily lifestyle behaviors.

INTERVENTIONS:
Behavioral: Exercise Training — Supervised exercise training
  Arms: CLL-EX

SUMMARY:
PURPOSE: The purpose of the study is to determine the effects of 12-weeks of exercise training on physical reserve, as measured by aerobic capacity, strength and physical function, in patients with CLL. Further, it is our aim to assess relationships with changes in physical reserve and resilience to the patient's cancer, as measured by immune cell counts, tumor cell killing and antibacterial functions.

DESIGN: Subjects will have confirmed treatment naïve CLL. Subjects will be assigned to either a 12-week control (no supervised exercise) or an intervention (HIIT) group. Before and after the 12 week program subjects will undergo several tests including: 1) a maximal treadmill test, 2) body composition, 3) muscle strength and endurance, 4) physical activity levels, 5) blood measures (e.g. immune and inflammatory functions). Subjects in the HIIT group will complete a 12-week supervised exercise training program consisting of HIIT and strength training.

DATA ANALYSES & SAFETY ISSUES: This is a pilot study, with the goal of assessing whether exercise training causes a change in aerobic fitness (VO2peak), muscle function, and immunological measures. Vo2peak will be measured by a cardiopulmonary exercise test, muscle function will be measured by strength tests, and immunological functions will be measured from blood samples. For outcomes, group change differences from baseline to 12-weeks will be compared by ANCOVA. The data will be used to provide power calculations for future grant proposals. High Intensity Interval Training is a very safe exercise modality. The regular use of vigorous intensity exercise intervals have been used extensively in exercise training. In fact, the exercise intervals will start at levels lower and will be of shorter duration than were used during the maximal exercise test. They will then be carefully and slowly made to be more challenging as each subject is able to safely tolerate.

HYPOTHESIS: The investigators hypothesize that HIIT will be a feasible exercise intervention for people with CLL and will result in improvements in markers of health and fitness.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CLL as per the International Workshop on CLL Guidelines.
* Male or female ≥ 18 years of age
* No history of prior treatment of CLL
* Able to walk on a treadmill or cycle on an ergometer
* Pass the CPET evaluation of aerobic fitness and cardiac health

Exclusion Criteria:

* Clinical evidence of significant disease progression with first line therapy expected within 6 months
* Corticosteroid therapy initiated less than 7 days prior to study entry. Prednisone 10mg or less or equivalent is allowed as clinically warranted. Topical or inhaled corticosteroids are permitted.
* Malignancy within 3 years of study enrollment requiring intervention except for adequately treated basal, squamous cell carcinoma or non-melanomatous skin cancer, carcinoma in situ of the cervix, superficial bladder cancer not treated with intravesical chemotherapy or BCG within 6 months, localized prostate cancer and PSA stable
* Absolute contra-indications to exercise: Recent (<6 months) acute cardiac event unstable angina, uncontrolled dysrhythmias causing symptoms or hemodynamic compromise, symptomatic aortic stenosis, uncontrolled symptomatic heart failure, acute pulmonary embolus, acute myocarditis or pericarditis, suspected or known dissecting aneurism and acute systemic infection.
* Significant orthopedic limitations, musculoskeletal disease and/or injury. Due to the nature of the study, persons with known joint, muscle or other orthopedic limitations that restrict physical activity may be excluded.
* Type I diabetes mellitus or uncontrolled Type II diabetes mellitus (HbA1c >7%), or chronic obstructive pulmonary disease
* Uncontrolled blood pressure (≥180/90) at rest during screening and confirmed on repeat manual measurement
* Unable to travel to fitness center or comply with other study requirements
* Known concurrent HIV, Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Change in VO2peak as measured by cardiopulmonary exercise test | Baseline to 12-weeks

SECONDARY OUTCOMES:
Change in lymphocyte doubling rate (LDR) as measured by blood test | Baseline to 12-weeks
Change in muscle strength as measured by a strength test | Baseline to 12-weeks
  Strength test is the estimated maximal amount of weight a subject can lift
Change in muscle endurance as measured by a muscle endurance test | Baseline to 12-weeks
  Endurance test is the amount of times a subject can lift 70% of maximal muscle strength
Change in neutrophil to lymphocyte ratio (NLR) as measured by blood test | Baseline to 12-weeks
Change in lymphocyte to monocyte ratio (LMR) as measured by blood test | Baseline to 12-weeks
Change in natural killer cell killing of tumor cell lines as measured by flow cytometry | Baseline to 12-weeks
Change in neutrophil killing of E.coli as measured by flow cytometry | Baseline to 12-weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Bartlett, PhD, Principal Investigator — Duke University; Andrea Sitlinger, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Artese AL, Sitlinger A, MacDonald G, Deal MA, Hanson ED, Pieper CF, Weinberg JB, Brander DM, Bartlett DB. Effects of high-intensity interval training on health-related quality of life in chronic lymphocytic leukemia: A pilot study. J Geriatr Oncol. 2023 Jan;14(1):101373. doi: 10.1016/j.jgo.2022.09.002. Epub 2022 Sep 9. PMID 36096873
- [Derived] MacDonald G, Sitlinger A, Deal MA, Hanson ED, Ferraro S, Pieper CF, Weinberg JB, Brander DM, Bartlett DB. A pilot study of high-intensity interval training in older adults with treatment naive chronic lymphocytic leukemia. Sci Rep. 2021 Nov 30;11(1):23137. doi: 10.1038/s41598-021-02352-6. PMID 34848750